CLINICAL TRIAL: NCT04056845
Title: Prospective Randomized Study on the Effects of Valgus Knee Brace for Knee Osteoarthritis in Chinese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Keith Hay-Man Wan, Resident Specialist, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HAREC
Record Dates: First submitted 2019-05-29; First posted 2019-08-14 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities; Analgesics; Diclofenac; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors are blinded from the treatment received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee brace group (Experimental): Patients in this group will receive a valgus knee brace (Medex K39-OA Corrector), to be worn for at least four hours a day, during the study period, on top of the presrciption of physiotherapy and oral analgesic (diclofenac and panadol).
  Interventions: Device: Valgus knee brace (Medex K39-OA Corrector); Other: Physiotherapy and oral analgesic (diclofenac and panadol)
- Control Group (Active Comparator): Patients in this group will receive physiotherapy and oral analgesic (diclofenac and panadol).
  Interventions: Other: Physiotherapy and oral analgesic (diclofenac and panadol)

INTERVENTIONS:
Device: Valgus knee brace (Medex K39-OA Corrector) — Valgus knee brace given to patients as part of the conservative management for knee osteoarthritis.
  Arms: Knee brace group
Other: Physiotherapy and oral analgesic (diclofenac and panadol) — Physiotherapy and oral analgesic (diclofenac and panadol)

SUMMARY:
To investigate whether the use of valgus knee brace is useful for patients with medial knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis of the knee is the commonest type of arthritis affecting both the middle age and geriatric population, which poses a huge burden to our in-patient and out-patient orthopaedic services. Conservative treatment like physiotherapy and analgesic provide temporary symptomatic relief. Surgical treatment like high tibial osteotomy and knee arthroplasty are not without major potential surgical risks and implant-related complications.

Orthotic treatment can theoretically alter the loading to the knee joint and help to reduce the symptoms and disease progression. Small scale biomechanical studies have demonstrated such effects with the use of valgus knee brace (2-4). Though prospective clinical outcome studies on Chinese patients in our locality are lacking.

Valgus knee brace is a non-pharmaceutical, non-invasive option for knee pain. Using a three-point leverage the unloader brace is to shift the stress away from the arthritic area to the normal portion of the knee, maintains good alignment and stability and thus provides significant pain relief during daily activities. It has been commonly used as a first line management option in other countries.

Our aim is to perform a prospective randomized study to look at the difference in outcome measures in osteoarthritic patients with the use of valgus knee brace, on top of the usual regime of conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-80
* History of symptomatic medial unicompartmental knee osteoarthritis > 6 months
* Willingness to wear the knee brace for a minimum of 4 hours per day during daily activities
* Understanding of the Chinese language
* Ethnic Chinese patients

Exclusion Criteria:

* Symptomatic knee osteoarthritis affecting more than one compartment
* Clinical and radiological signs of osteoarthritis over the lateral compartment or patello-femoral joint
* Significant knee effusion or soft tissue compromise preventing long-term knee brace use
* Obesity (BMI>30)
* Previous surgery on the affected knee other than diagnostic arthroscopy with debridement, soft tissue reconstruction, menisectomy
* Peripheral vascular disease of the lower limb

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in pain | At 16 weeks after the initiation of study
  Visual Analog Scale (VAS) for pain from 0 to 10, with higher value signifying worse pain control

SECONDARY OUTCOMES:
Improvement in knee functioning | At 16 weeks after the initiation of the study
  The Western Ontario and McMaster Universities Osteoarthritis Index

CONTACTS AND LOCATIONS:
Overall Officials: Keith Hay-Man Wan, MBChB, FRCSEd(Orth), Principal Investigator — Hospital Authority
Locations (1):
- Hospital Authority, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu HC, Lie CW, Ng TP, Chen KW, Tse CY, Wong WH. Prospective study on the effects of orthotic treatment for medial knee osteoarthritis in Chinese patients: clinical outcome and gait analysis. Hong Kong Med J. 2015 Apr;21(2):98-106. doi: 10.12809/hkmj144311. Epub 2015 Mar 10. PMID 25756275
- [Background] Moyer RF, Birmingham TB, Bryant DM, Giffin JR, Marriott KA, Leitch KM. Valgus bracing for knee osteoarthritis: a meta-analysis of randomized trials. Arthritis Care Res (Hoboken). 2015 Apr;67(4):493-501. doi: 10.1002/acr.22472. PMID 25201520

DOCUMENTS (1):
  • Study Protocol (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT04056845/Prot_002.pdf